CLINICAL TRIAL: NCT07134946
Title: In Vitro Study on Donor Corneas Preservation in IRESTORE Storage Medium. A Post Marketing Interventional Study on Device
Acronym: IRESTORE
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Roberto Ceccuzzi, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: IRESTORE storage medium
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Donor Corneas Preservation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Donor corneas are harvested and then stored in the Eye Bank to maintain their viability until analysis and subsequent release for transplantation. The storage period of donor corneas is classified in terms of duration and storage temperature: short-intermediate cold (up to two weeks between 2 and 6°C) and long-term warm (up to 4 weeks between 31 and 37°C). Corneal tissues are initially collected and stored cold at 4°C. After evaluation they can be stored in cold storage medium until transplantation or placed in organ culture at 31°C. IRESTORE, a cold storage liquid, has recently become available.

DETAILED DESCRIPTION:
The device used in the study is classified as class II A (medium risk) The device iRestore Conservation, sterile liquid for the preservation of corneal grafts in hypothermic conditions up to 14 days. Consists of a 20 ml solution suitable for the temporary preservation of corneal tissues in hypothermia split into a cylindric, optical bottom glass vial, which provides specular microscope examination.

It contains dextran as Osmotic agent; sodium pyruvate, glucose as energy source; salts, aminoacids, vitamins as nutritional sources; gentamycin: 143 µg/mL as preservative system; HEPES, sodium bicarbonate as pH Buffer; Phenol red as pH indicator.

ELIGIBILITY:
Inclusion criteria (donor):

* Medical history of a disease that excludes donation;
* serological positivity (HBV, HCV, HIV);

Inclusion criteria (cornea):

* low endothelial cell density (<2000 cells/mm2);
* stromal opacities.

Exclusion criteria (cornea):

* Severe endothelial dystrophy;
* massive endothelial mortality;
* marked stromal opacities.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: donor corneas
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-11-07 (Estimated); Study Completion 2025-11-07 (Estimated)

PRIMARY OUTCOMES:
cell density | 7 days
  endothelial cell density at day 7

SECONDARY OUTCOMES:
cell density over time | days 1, 3, 7, 10, 14
  Change of corneal transparency, endothelial cell density, polymorphism (hexagonality), polymegatism, and pachymetry as a function of storage time of endothelial cells over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy